CLINICAL TRIAL: NCT03252574
Title: To Explore the Physiological Impact of AIR+ Smart Masks on Children
Brief Title: A Randomised Crossover Study to Explore the Physiological Impact of AIR+ Smart Masks on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innosparks Pte Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other); KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ISPL-2015/01059
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence AB (Other): No mask, followed by AIR+ Smart Mask only (A), then AIR+ Smart Mask with micro-ventilator (B)
  Interventions: Other: A; Other: B
- Sequence BA (Other): No mask, followed by AIR+ Smart Mask with micro-ventilator (B), then AIR+ Smart Mask only (A).
  Interventions: Other: A; Other: B

INTERVENTIONS:
Other: A — AIR+ Smart Mask Only
Other: B — AIR+ Smart Mask with micro-ventilator

SUMMARY:
The primary objective is to evaluate the physiological impact of AIR+ Smart Masks on end-tidal carbon dioxide (ETCO2) of children aged 7 to 14 years of age. The secondary outcomes include other physiological parameters such as oxygen saturation (SPO2), heart rate (HR) and respiratory rate (RR). In addition, we will assess the general well-being and comfort level of the child when wearing the AIR+Smart Mask with and without micro-ventilator.

DETAILED DESCRIPTION:
Studies have shown that prolonged wearing of disposable particulate respirators may lead to an increase in carbon dioxide (CO2) levels in the dead space of the respirator as well as in the re-breathing of the expired air when wearing it. The increased CO2 levels may result in headaches, increased irritability, and breathing difficulty. In addition, there is some discomfort due to the accumulation of heat and humid air in the dead space of between the respirator and face. Innosparks Pte Ltd (formerly, ST Dynamics) (the Advanced Engineering Centre of ST Engineering) developed a new type of disposable particulate respirator (hereon referred to as AIR+ Smart Mask) that is suitable for use in both adults and children, from ages 7 and above.They also designed an optional accompanying device, the micro-ventilator, which is battery-powered and aims to extract accumulated heat, moisture, and carbon dioxide from within the mask. Innosparks Pte Ltd (formerly, ST Dynamics) have obtained the US National Institute for Occupational Safety and Health (NIOSH) N95 certification for the three sizes of masks without micro-ventilator, and Conformité Européenne's (CE) certification for the following mask specifications:• FFP1 and NIOSH approved N95 for S and M-sized AIR+ Smart Masks without micro ventilator;• FFP2 and NIOSH approved N95 for L-sized mask without micro ventilator;• FFP1 certification for S and M-sized masks with micro-ventilator, and;• FFP2 certification for the L size mask with micro-ventilator.For purposes of this research, both CE and NIOSH markings will be made for the masks trialed.As the masks were developed specifically for school-going children, this study is designed to explore whether the new disposable particulate respirator, which can be attached with a ventilator to vent out expired air within the respirator, is safe and effective for use in healthy children aged 7 to 14 years of age. This is through measuring the variation of carbon dioxide levels in children with and without the AIR+ Smart Mask. End-tidal carbon dioxide pressure (ETCO2) is a good indicator of arterial carbon dioxide pressure (PaCO2) in healthy adults and children, and has been used for continuous direct assessment of PaCO2 in clinical contexts. The normal range of PaCO2 is from 35 - 45 mmHg. As there is a slight margin of difference between ETCO2 and PaCO2 values during measurement of about 1.6 +/- 4.3mmHg, this study defines 30 to 50mmHg as the acceptable range for ETCO2 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 7 and 14 years of age (inclusive)
2. Subjects and their parent/legal guardian must provide the consent and assent as appropriate to take part in this study.

Exclusion Criteria:

1. Subjects with any known cardiorespiratory conditions (including but not limited to the following: asthma, bronchitis, cystic fibrosis, congenital heart disease, emphysema)
2. Subjects with any known medical conditions that may be exacerbated by strenuous activity, including but not limited to the following: exercise-induced asthma, lower respiratory infection (including pneumonia, bronchitis) in the past 2 weeks, anxiety disorders, diabetes, hypertension, or epilepsy/ seizure disorder
3. Subjects with any physical disability from medical, orthopaedic or neuromuscular disorders
4. Subjects who have an acute upper respiratory tract infection/ moderately severe rhinitis (i.e. blocked nasal passages) on the day of the study
5. Subjects who may compromise the integrity of the mask fit (e.g. those with excessive facial hair).

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2016-07; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
End Tidal Carbon Dioxide | 75 minutes

SECONDARY OUTCOMES:
Percent Oxygen Saturation | 75 minutes
Heart Rate | 75 minutes
Respiratory Rate | 75 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Goh, A/P, Principal Investigator — NUH
Locations (1):
- Innosparks Pte Ltd, 75 Ayer Rajah Crescent, #02-13, Singapore, Singapore

REFERENCES:
- [Background] Roberge RJ, Coca A, Williams WJ, Powell JB, Palmiero AJ. Physiological impact of the N95 filtering facepiece respirator on healthcare workers. Respir Care. 2010 May;55(5):569-77. PMID 20420727
- [Background] Sinkule EJ, Powell JB, Goss FL. Evaluation of N95 respirator use with a surgical mask cover: effects on breathing resistance and inhaled carbon dioxide. Ann Occup Hyg. 2013 Apr;57(3):384-98. doi: 10.1093/annhyg/mes068. Epub 2012 Oct 29. PMID 23108786
- [Background] Ickx B, Dolomie J-0, Benalouch M et al. Arterial to End-tidal carbon dioxide tension differences in infants and children, JACR, 2155-6148 6: 511. doi:10.4172/2155-6148.1000511